CLINICAL TRIAL: NCT00151125
Title: Phase II Comparison Study of Hemostatic Efficacy of Escalating Doses of Interleukin-11 (rhIL-11, Neumega) in Subjects With Type 1 Von Willebrand Disease
Brief Title: Phase II Study of IL-11 (Neumega) in Von Willebrand Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); University of North Carolina (Other)
Responsible Party: Principal Investigator, Margaret Ragni, Professor of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0403006; 0403006 (Other: protocol id)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Von Willebrand Disease
Keywords: Von Willebrand Disease; Bleeding; Coagulation; Hemostatic agent
MeSH Terms: conditions — von Willebrand Diseases; Hemorrhage; Thrombosis | interventions — Interleukin-11; oprelvekin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): rhIL-11 (Interleukin-11, Neumega) 25 mcg/kg subcutaneously daily for 7 days
  Interventions: Drug: recombinant interleukin-11
- B (Experimental): rhIL-11 (interleukin-11, Neumega) 50 mcg/kg subcutaneously daily for 7 days
  Interventions: Drug: recombinant interleukin-11
- C (Experimental): rhIL-11 (Interleukin-11, Neumega) 10 mg/kg subcutaneously daily for 7 days
  Interventions: Drug: recombinant interleukin-11

INTERVENTIONS:
Drug: recombinant interleukin-11 — 25 mcg/kg subcutaneously daily for seven days
  Other Names: rhIL-11, Neumega
  Arms: A
Drug: recombinant interleukin-11 — 50 mcg/kg subcutaneously daily for 7 days
  Other Names: rhIL-11, Neumega
  Arms: B
Drug: recombinant interleukin-11 — 10 mcg/kg subcutaneously daily for 7 days
  Other Names: rhIL-11, Neumega
  Arms: C

SUMMARY:
This study is testing the use of rhIL-11 (recombinant interleukin 11, Neumega) in individuals with Von Willebrand disease. The purpose is to evaluate:

1. if rhIL-11 corrects VWF (Von Willebrand Factor) levels to normal
2. if rhIL-11 and DDAVP together will boost VWF levels even higher
3. the onset, peak, and duration of rhIL-11 effect
4. if rhIL-11 is safe in individuals with Von Willebrand Disease

DETAILED DESCRIPTION:
This is a prospective, single center, open-label, escalating dose Phase II comparison study of interleukin-11 (rhIL-11, Neumega) in subjects with type 1 Von Willebrand Disease (VWD).

The purpose is to establish the clinical safety and hemostatic efficacy of rhIL-11 in individuals with type 1 Von Willebrand disease.

Study subjects will include the following subjects:

1. age >= 18 years of age
2. diagnosis of VWD confirmed by: 2a) at least 2 of 4 abnormal vWD-related coagulation tests; 2b) a past bleeding history

A total of 10-16 subjects are anticipated to be enrolled and complete the study. The specific aims of the study are:

1. to compare the hemostatic efficacy of three escalating doses of rhIL-11
2. to determine the biologic effects of rhIL-11
3. to determine whether DDAVP, when given after the seventh daily dose of rhIL-11, enhances hemostatic efficacy or rhIL-11
4. to compare the safety of three escalating doses of rhIL-11

Efficacy will be based on the number and percent increase of VWD-related coagulation tests into the normal range, or at least to 2-3 times baseline.

Safety will be based on the number and frequency of adverse reactions, including fever, headache, fatigue, arthralgias, myalgias, fluid retention, and edema.

The study will last up to 4 weeks per subject, and for 24 months for the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older
* Confirmed VWD by 2 of 4 VWD coagulation tests abnormal
* A past bleeding history
* No hormone, oral contraceptive, estrogen use in past 8 weeks
* Willingness to have blood drawn
* Willingness to sign informed consent

Exclusion Criteria:

* Presence of other bleeding disorder, e.g. acquired VWD, thrombocytopenia
* Use of estrogens, hormones, oral contraceptives in past 8 weeks
* Use of immunomodulatory or experimental drugs or diuretics
* Pregnant or lactating women
* Past cardiac disease, congestive failure, arrhythmia (e.g. atrial fibrillation, atrial flutter), hypertension, MI, stroke, or thrombosis
* Past allergic reaction to Neumega or DDAVP
* Surgery within the past 8 weeks
* Inability to comply with study protocol requirements
* Concomitant use of antiplatelet drugs, anticoagulants, dextran, aspirin, or NSAIDs
* Treatment with DDAVP, cryoprecipitate, whole blood, plasma, and plasma derivatives containing FVIII, VWF within 5 days of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The number and percent increase of VWD coagulation tests after seven daily doses of rhIL-11, boosted by DDAVP day 7. | The time frame is up to 14 days per subject.

SECONDARY OUTCOMES:
The number and frequency of IL-11 associated adverse events. | The time frame is up to 14 days per subject.
The mechanism of IL-11 biologic effect by VWFmRNA. | The time frame is within 14 days per subject.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V. Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Hemophilia Center of Western Pennsylvania and General Clinical Research Center, Pittsburgh, Pennsylvania, United States